CLINICAL TRIAL: NCT02485301
Title: Safety and Immunogenicity Study of GSK Biologicals' Investigational Recombinant Chimpanzee Adenovirus Type 3-vectored Ebola Zaire Vaccine (GSK3390107A) in Adults in Africa
Brief Title: A Study to Evaluate the Safety and Immunogenicity of a Candidate Ebola Vaccine in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 202091
Record Dates: First submitted 2015-06-18; First posted 2015-06-30 (Estimated); Results first posted 2018-01-04 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2017-11

CONDITIONS: Virus Diseases
Keywords: Protection against Ebola Zaire virus
MeSH Terms: conditions — Virus Diseases | interventions — halofantrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group EBO-Z (Experimental): The subjects in the Group EBO-Z will receive the vaccine at Day 0 of the study
  Interventions: Biological: GlaxoSmithKline (GSK) Biologicals' investigational recombinant chimpanzee adenovirus Type 3-vectored Ebola Zaire vaccine (ChAd3-EBO-Z) (GSK3390107A)
- Group Placebo/ EBO-Z (Placebo Comparator): The subjects in the Group Placebo/ EBO-Z will receive a placebo at Day 0 (as a control) and will receive the investigational ChAd3-EBO-Z vaccine at Month 6
  Interventions: Biological: GlaxoSmithKline (GSK) Biologicals' investigational recombinant chimpanzee adenovirus Type 3-vectored Ebola Zaire vaccine (ChAd3-EBO-Z) (GSK3390107A); Drug: Placebo

INTERVENTIONS:
Biological: GlaxoSmithKline (GSK) Biologicals' investigational recombinant chimpanzee adenovirus Type 3-vectored Ebola Zaire vaccine (ChAd3-EBO-Z) (GSK3390107A) — A single dose administrated intramuscular
Drug: Placebo — A single dose administrated intramuscular
  Arms: Group Placebo/ EBO-Z

SUMMARY:
The purpose of this study is to assess the safety and immunogenicity of the investigational ChAd3-EBO-Z vaccine administered to approximately 3 000 adults in Africa as a single IM dose Considering the risk of exposure to Ebola and the potential (based on animal data) for the investigational ChAd3-EBO-Z vaccine to afford at least partial protection, all subjects in the study will receive the investigational ChAd3-EBO-Z vaccine. The subjects in the Group EBO-Z will receive the vaccine at Day 0 of the study, whereas the subjects in the Group Placebo/ EBO-Z will receive a placebo at Day 0 (as a control) and will receive the investigational ChAd3-EBO-Z vaccine at Month 6, provided that no safety concerns are raised. In addition, vaccinating all subjects in the study with the investigational ChAd3 EBO Z vaccine will allow an increase of the safety database of the investigational vaccine. In case the geographic range of Ebola virus Zaire (EBOV) transmission expands to encompass any of the regions where this trial is conducted, earlier administration of the investigational ChAd3-EBO-Z vaccine to the subjects in the Group Placebo/ EBO-Z will be considered in that region.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the Investigator, can and will comply with the requirements of the protocol (e.g. capability of or availability for Diary Card completion, return for follow-up visits, availability for clinical follow-up throughout the study period).
* Written/ thumb printed informed consent obtained from the subject prior to performing any study specific procedure or written/ thumb printed informed consent obtained from the subject's parent(s)/ legally acceptable representative(s) (LAR[s]) and written/ thumb printed informed assent obtained from the subject, for minor subjects. This will only be applicable for countries where the legal age of majority is ≥ 21 years.
* A male or female aged 18 years of age or older at the time of Screening.
* Healthy subjects as per Investigator judgement, as established by medical history, clinical examination and haematology/ biochemistry laboratory parameters screening before entering into the study.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:
* has practiced adequate contraception for 30 days prior to the Day 0 visit, and
* has a negative pregnancy test at the Day 0 visit, and
* has agreed to continue adequate contraception until 30 days after the Month 6 visit.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine during the period starting 30 days before the Day 0 visit, or planned use during the study period.
* Previous vaccination with an investigational EBOV or Marburg vaccine, or previous vaccination with a chimpanzee adenoviral vectored investigational vaccine.
* Known prior EBOV or SUDV disease.
* Travel to a country affected by the EBOV epidemic or direct contact with a person with EVD within 21 days prior to the Day 0 visit.
* History of any reaction or hypersensitivity (such as anaphylaxis, urticaria [hives], respiratory difficulty, angioedema, or abdominal pain) likely to be exacerbated by any component of the study vaccine.
* Planned administration/ administration of a vaccine not foreseen by the study protocol in the period starting 30 days before and ending 30 days after each vaccination visit.
* Serious acute or chronic illness determined by medical history and clinical examination including, but not limited to:

  * Clinically significant immunosuppressive or immunodeficient condition (e.g. clinical acquired immune deficiency syndrome [AIDS]).
  * Any clinically significant haematological (CBC, including differential count and platelet count) or biochemical (ALT, creatinine) laboratory abnormality.
  * Any chronic illness with recent signs of exacerbation, or imposing a change in the chronic treatment regimen, within 3 months prior to the Day 0 visit.
  * Any unstable chronic medical condition (e.g. uncontrolled asthma).
* Pregnant female.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3024 (Actual)
Dates: Start 2015-07-15 (Actual); Primary Completion 2016-12-23 (Actual); Study Completion 2016-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Cameroon (2):
  - GSK Investigational Site, Bamenda
  - GSK Investigational Site, Yaoundé
- GSK Investigational Site, Bamako, Mali
- GSK Investigational Site, Abuja, Nigeria
- GSK Investigational Site, Dakar, Senegal

REFERENCES:
- [Derived] Tapia MD, Sow SO, Ndiaye BP, Mbaye KD, Thiongane A, Ndour CT, Mboup S, Ake JA, Keshinro B, Akintunde GA, Kinge TN, Vernet G, Bigna JJ, Oguche S, Koram KA, Asante KP, Hogrefe WR, Gunther S, Naficy A, De Ryck I, Debois M, Bourguignon P, Jongert E, Ballou WR, Koutsoukos M, Roman F; Zaire EBola Research Alliance group. Safety, reactogenicity, and immunogenicity of a chimpanzee adenovirus vectored Ebola vaccine in adults in Africa: a randomised, observer-blind, placebo-controlled, phase 2 trial. Lancet Infect Dis. 2020 Jun;20(6):707-718. doi: 10.1016/S1473-3099(20)30016-5. Epub 2020 Mar 19. PMID 32199491

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening period the following steps took place: signing of informed consent, checking of inclusion/exclusion criteria, demographic data collection, medical history collection, physical examination, pregnancy testing.
Groups:
- GSK3390107A Group: Healthy male or female subjects, aged 18 or older at the time of screening, who received one dose of the investigational GSK3390107A vaccine, at Day 0, administered intramuscularly, into the deltoid region of the arm.
- Placebo+GSK3390107A Group: Healthy male or female subjects, aged 18 or older at the time of screening, who received one dose of placebo at Day 0 and one dose of the investigational GSK3390107A vaccine at Month 6, administered intramuscularly, into the deltoid region of the arm.
Period: Overall Study
Arm/Group | GSK3390107A Group | Placebo+GSK3390107A Group
Started (Out of 3024 subjects originally enrolled, only 3013 subjects received vaccination.) | 1509 | 1504
Completed | 1471 | 1455
Not Completed | 38 | 49
Not completed — Serious Adverse Events | 2 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 6 | 7
Not completed — Migrated/moved from study area | 10 | 19
Not completed — Lost to Follow-up | 17 | 17
Not completed — Other | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK3390107A Group | Placebo+GSK3390107A Group | Total
Number analyzed (Participants) | 1509 | 1504 | 3013
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.4 (12.71) | 33.0 (12.43) | 32.7 (12.57)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 697 | 690 | 1387
  Male | 812 | 814 | 1626
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: African heritage/African American | 1505 | 1501 | 3006
  Geographic ancestry: American Indian or Alaskan native | 1 | 0 | 1
  Geographic ancestry: Asian - Japanese heritage | 1 | 0 | 1
  Geographic ancestry: Asian - South East Asian heritage | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Solicited Local Adverse Events
Description: Assessed solicited local adverse events were pain, redness and swelling. Any = occurrence of any solicited local adverse event regardless of their intensity grade. Grade 3 Pain = significant pain at rest. Prevented normal every day activities. Grade 3 Redness/Swelling = redness/swelling spreading beyond 100 millimeters (mm) from injection site.
Time Frame: During the 7-Day (Days 0-6) post-vaccination period
Population: The analysis was performed on the Total Vaccinated Cohort - Adverse Event (AE) and Humoral Immunity Sub-cohort, which included all subjects with at least one vaccine administration documented, who filled in their symptom sheets.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3390107A Group | Placebo+GSK3390107A Group
Number analyzed (Participants) | 748 | 751
Participants
  Any Pain | 356 | 57
  Grade 3 Pain | 3 | 0
  Any Redness | 2 | 0
  Grade 3 Redness | 0 | 0
  Any Swelling | 9 | 5
  Grade 3 Swelling | 0 | 0

2. Primary Outcome: Number of Subjects With Solicited General Adverse Events
Description: Assessed solicited general adverse events were fatigue, fever [defined as axillary temperature higher than or equal to (≥) 37.5 degrees Celsius (°C)], gastrointestinal (gastro) adverse events [nausea, vomiting, diarrhoea and/or abdominal pain] and headache. Any = occurrence of any general adverse events regardless of intensity grade or relationship to vaccination. Grade 3 fatigue, gastrointestinal symptoms and headache = adverse event that prevented normal activities. Grade 3 fever = fever ≥ 39.5 °C. Related = adverse event assessed by the investigator as related to the vaccination.
Time Frame: During the 7-Day (Days 0-6) post-vaccination period
Population: The analysis was performed on the Total Vaccinated Cohort - AE and Humoral Immunity Sub-cohort, which included all subjects with at least one vaccine administration documented, who filled in their symptom sheets.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3390107A Group | Placebo+GSK3390107A Group
Number analyzed (Participants) | 748 | 751
Participants
  Any Fatigue | 284 | 94
  Grade 3 Fatigue | 11 | 3
  Related Fatigue | 243 | 72
  Any Fever | 106 | 24
  Grade 3 Fever | 3 | 0
  Related Fever | 88 | 17
  Any Gastro | 73 | 49
  Grade 3 Gastro | 2 | 0
  Related Gastro | 57 | 40
  Any Headache | 345 | 136
  Grade 3 Headache | 10 | 4
  Related Headache | 306 | 104

3. Primary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset out-side the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 30-Day (Days 0-29) post-vaccination period
Population: The analysis was performed on the Total Vaccinated Cohort - AE and Humoral Immunity Sub-cohort, which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3390107A Group | Placebo+GSK3390107A Group
Number analyzed (Participants) | 749 | 751
Participants | 123 | 119

4. Primary Outcome: Percentage of Subjects With Haematological Laboratory Abnormalities
Description: Haematological parameters assessed included: complete blood count (red blood cells [RBC], neutrophils, lymphocytes, white blood cells [WBC], haemoglobin), as well as differential count and platelet count. Reference range indicators used were: high, low, normal.
Time Frame: At Screening
Population: The analysis was performed on the Total Vaccinated Cohort - AE and Humoral Immunity Sub-cohort, which included all subjects with at least one vaccine administration documented and with available results at Screening.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A Group | Placebo+GSK3390107A Group
Number analyzed (Participants) | 665 | 667
Percentage of participants
  RBC, Low | 14.6 | 14.2
  RBC, Normal | 70.8 | 69.1
  RBC, High | 14.6 | 16.6
  Neutrophils, Low: number analyzed (Participants) | 588 | 588
  Neutrophils, Low | 50.2 | 48.3
  Neutrophils, Normal: number analyzed (Participants) | 588 | 588
  Neutrophils, Normal | 49.5 | 51.5
  Neutrophils, High: number analyzed (Participants) | 588 | 588
  Neutrophils, High | 0.3 | 0.2
  Lymphocytes, Low: number analyzed (Participants) | 588 | 588
  Lymphocytes, Low | 0.9 | 1.0
  Lymphocytes, Normal: number analyzed (Participants) | 588 | 588
  Lymphocytes, Normal | 97.8 | 98.0
  Lymphocytes, High: number analyzed (Participants) | 588 | 588
  Lymphocytes, High | 1.4 | 1.0
  WBC, Low | 9.3 | 8.7
  WBC, Normal | 88.6 | 89.7
  WBC, High | 2.1 | 1.6
  Haemoglobin, Low | 17.6 | 18.1
  Haemoglobin, Normal | 80.6 | 79.5
  Haemoglobin, High | 1.8 | 2.4
  Platelets, Low | 2.9 | 1.8
  Platelets, Normal | 90.4 | 92.5
  Platelets, High | 6.8 | 5.7

5. Primary Outcome: Percentage of Subjects With Haematological Laboratory Abnormalities
Description: as for outcome 4
Time Frame: At Day 3
Population: The analysis was performed on the Total Vaccinated Cohort - AE and Humoral Immunity Sub-cohort, which included all subjects with at least one vaccine administration documented and with available results at Day 3.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A Group | Placebo+GSK3390107A Group
Number analyzed (Participants) | 659 | 662
Percentage of participants
  RBC, Low | 19.0 | 20.4
  RBC, Normal | 70.9 | 66.5
  RBC, High | 10.2 | 13.1
  Neutrophils, Low: number analyzed (Participants) | 583 | 583
  Neutrophils, Low | 77.9 | 56.8
  Neutrophils, Normal: number analyzed (Participants) | 583 | 583
  Neutrophils, Normal | 21.8 | 42.7
  Neutrophils, High: number analyzed (Participants) | 583 | 583
  Neutrophils, High | 0.3 | 0.5
  Lymphocytes, Low: number analyzed (Participants) | 583 | 583
  Lymphocytes, Low | 2.9 | 1.4
  Lymphocytes, Normal: number analyzed (Participants) | 583 | 583
  Lymphocytes, Normal | 96.4 | 97.8
  Lymphocytes, High: number analyzed (Participants) | 583 | 583
  Lymphocytes, High | 0.7 | 0.9
  WBC, Low | 17.9 | 10.7
  WBC, Normal | 80.7 | 87.8
  WBC, High | 1.4 | 1.5
  Haemoglobin, Low | 25.9 | 27.0
  Haemoglobin, Normal | 72.5 | 72.2
  Haemoglobin, High | 1.5 | 0.8
  Platelets, Low | 2.3 | 2.3
  Platelets, Normal | 94.1 | 91.8
  Platelets, High | 3.6 | 5.9

6. Primary Outcome: Percentage of Subjects With Haematological Laboratory Abnormalities
Description: as for outcome 4
Time Frame: At Day 6
Population: The analysis was performed on the Total Vaccinated Cohort - AE and Humoral Immunity Sub-cohort, which included all subjects with at least one vaccine administration documented and with available results at Day 6.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A Group | Placebo+GSK3390107A Group
Number analyzed (Participants) | 659 | 664
Percentage of participants
  RBC, Low | 20.6 | 21.5
  RBC, Normal | 68.6 | 67.2
  RBC, High | 10.8 | 11.3
  Neutrophils, Low: number analyzed (Participants) | 584 | 585
  Neutrophils, Low | 65.2 | 53.5
  Neutrophils, Normal: number analyzed (Participants) | 584 | 585
  Neutrophils, Normal | 34.2 | 46.2
  Neutrophils, High: number analyzed (Participants) | 584 | 585
  Neutrophils, High | 0.5 | 0.3
  Lymphocytes, Low: number analyzed (Participants) | 584 | 585
  Lymphocytes, Low | 0.9 | 2.4
  Lymphocytes, Normal: number analyzed (Participants) | 584 | 585
  Lymphocytes, Normal | 97.8 | 96.2
  Lymphocytes, High: number analyzed (Participants) | 584 | 585
  Lymphocytes, High | 1.4 | 1.4
  WBC, Low | 14.7 | 10.7
  WBC, Normal | 83.5 | 87.7
  WBC, High | 1.8 | 1.7
  Haemoglobin, Low | 28.2 | 27.4
  Haemoglobin, Normal | 71.3 | 72.0
  Haemoglobin, High | 0.5 | 0.6
  Platelets, Low | 2.4 | 2.0
  Platelets, Normal | 91.5 | 91.9
  Platelets, High | 6.1 | 6.2

7. Primary Outcome: Percentage of Subjects With Haematological Laboratory Abnormalities
Description: as for outcome 4
Time Frame: At Day 30
Population: The analysis was performed on the Total Vaccinated Cohort - AE and Humoral Immunity Sub-cohort, which included all subjects with at least one vaccine administration documented and with available results at Day 30.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A Group | Placebo+GSK3390107A Group
Number analyzed (Participants) | 658 | 661
Percentage of participants
  RBC, Low | 15.8 | 17.4
  RBC, Normal | 67.0 | 67.6
  RBC, High | 17.2 | 15.0
  Neutrophils, Low: number analyzed (Participants) | 583 | 583
  Neutrophils, Low | 56.4 | 55.6
  Neutrophils, Normal: number analyzed (Participants) | 583 | 583
  Neutrophils, Normal | 43.6 | 43.7
  Neutrophils, High: number analyzed (Participants) | 583 | 583
  Neutrophils, High | 0 | 0.7
  Lymphocytes, Low: number analyzed (Participants) | 583 | 583
  Lymphocytes, Low | 2.4 | 2.2
  Lymphocytes, Normal: number analyzed (Participants) | 583 | 583
  Lymphocytes, Normal | 96.2 | 97.3
  Lymphocytes, High: number analyzed (Participants) | 583 | 583
  Lymphocytes, High | 1.4 | 0.5
  WBC, Low | 12.3 | 12.1
  WBC, Normal | 86.8 | 86.5
  WBC, High | 0.9 | 1.4
  Haemoglobin, High | 23.4 | 23.0
  Haemoglobin, Normal | 75.4 | 75.8
  Haemoglobin, Low | 1.2 | 1.2
  Platelets, Low | 3.3 | 2.3
  Platelets, Normal | 92.6 | 91.5
  Platelets, High | 4.1 | 6.2

8. Primary Outcome: Percentage of Subjects With Haematological Laboratory Abnormalities
Description: as for outcome 4
Time Frame: At Month 6
Population: The analysis was performed on the Total Vaccinated Cohort - AE and Humoral Immunity Sub-cohort, which included all subjects with at least one vaccine administration documented and with available results at Month 6.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A Group | Placebo+GSK3390107A Group
Number analyzed (Participants) | 649 | 645
Percentage of participants
  RBC, Low | 16.2 | 17.2
  RBC, Normal | 69.5 | 67.9
  RBC, High | 14.3 | 14.9
  Neutrophils, Low: number analyzed (Participants) | 574 | 572
  Neutrophils, Low | 50.9 | 50.2
  Neutrophils, Normal: number analyzed (Participants) | 574 | 572
  Neutrophils, Normal | 48.6 | 49.5
  Neutrophils, High: number analyzed (Participants) | 574 | 572
  Neutrophils, High | 0.5 | 0.3
  Lymphocytes, Low: number analyzed (Participants) | 574 | 572
  Lymphocytes, Low | 1.7 | 1.6
  Lymphocytes, Normal: number analyzed (Participants) | 574 | 572
  Lymphocytes, Normal | 96.9 | 97.4
  Lymphocytes, High: number analyzed (Participants) | 574 | 572
  Lymphocytes, High | 1.4 | 1.0
  WBC, Low | 13.3 | 10.9
  WBC, Normal | 85.4 | 88.2
  WBC, High | 1.4 | 0.9
  Haemoglobin, Low | 30.5 | 29.0
  Haemoglobin, Normal | 68.7 | 70.1
  Haemoglobin, High | 0.8 | 0.9
  Platelets, Low | 2.6 | 2.0
  Platelets, Normal | 93.2 | 94.6
  Platelets, High | 4.2 | 3.4

9. Primary Outcome: Percentage of Subjects With Haematological Laboratory Abnormalities
Description: as for outcome 4
Time Frame: At Month 6 + 6 Days
Population: The analysis was performed on the Total Vaccinated Cohort - AE and Humoral Immunity Sub-cohort, which included all subjects with at least one vaccine administration documented and with available results at Month 6 + 6 Days timepoint.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A Group | Placebo+GSK3390107A Group
Number analyzed (Participants) | 0 | 619
Percentage of participants
  RBC, Low |  | 18.6
  RBC, Normal |  | 70.1
  RBC, High |  | 11.3
  Neutrophils, Low: number analyzed (Participants) | 0 | 549
  Neutrophils, Low |  | 57.4
  Neutrophils, Normal: number analyzed (Participants) | 0 | 549
  Neutrophils, Normal |  | 42.4
  Neutrophils, High: number analyzed (Participants) | 0 | 549
  Neutrophils, High |  | 0.2
  Lymphocytes, Low: number analyzed (Participants) | 0 | 549
  Lymphocytes, Low |  | 0.7
  Lymphocytes, Normal: number analyzed (Participants) | 0 | 549
  Lymphocytes, Normal |  | 97.8
  Lymphocytes, High: number analyzed (Participants) | 0 | 549
  Lymphocytes, High |  | 1.5
  WBC, Low |  | 12.3
  WBC, Normal |  | 86.4
  WBC, High |  | 1.3
  Haemoglobin, Low |  | 36.3
  Haemoglobin, Normal |  | 63.2
  Haemoglobin, High |  | 0.5
  Platelets, Low |  | 1.8
  Platelets, Normal |  | 94.5
  Platelets, High |  | 3.7

10. Primary Outcome: Percentage of Subjects With Haematological Laboratory Abnormalities
Description: as for outcome 4
Time Frame: At Month 6 + 30 Days
Population: The analysis was performed on the Total Vaccinated Cohort - AE and Humoral Immunity Sub-cohort, which included all subjects with at least one vaccine administration documented and with available results at Month 6 + 30 Days timepoint.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A Group | Placebo+GSK3390107A Group
Number analyzed (Participants) | 0 | 616
Percentage of participants
  RBC, Low |  | 21.6
  RBC, Normal |  | 66.1
  RBC, High |  | 12.3
  Neutrophils, Low: number analyzed (Participants) | 0 | 547
  Neutrophils, Low |  | 55.9
  Neutrophils, Normal: number analyzed (Participants) | 0 | 547
  Neutrophils, Normal |  | 43.7
  Neutrophils, High: number analyzed (Participants) | 0 | 547
  Neutrophils, High |  | 0.4
  Lymphocytes, Low: number analyzed (Participants) | 0 | 547
  Lymphocytes, Low |  | 2.0
  Lymphocytes, Normal: number analyzed (Participants) | 0 | 547
  Lymphocytes, Normal |  | 96.3
  Lymphocytes, High: number analyzed (Participants) | 0 | 547
  Lymphocytes, High |  | 1.6
  WBC, Low |  | 11.4
  WBC, Normal |  | 87.7
  WBC, High |  | 1.0
  Haemoglobin, Low |  | 34.3
  Haemoglobin, Normal |  | 65.1
  Haemoglobin, High |  | 0.6
  Platelets, Low |  | 2.4
  Platelets, Normal |  | 94.6
  Platelets, High |  | 2.9

11. Primary Outcome: Percentage of Subjects With Haematological Laboratory Abnormalities
Description: as for outcome 4
Time Frame: At Month 12
Population: The analysis was performed on the Total Vaccinated Cohort - AE and Humoral Immunity Sub-cohort, which included all subjects with at least one vaccine administration documented and with available results at Month 12.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A Group | Placebo+GSK3390107A Group
Number analyzed (Participants) | 627 | 631
Percentage of participants
  RBC, Low | 15.3 | 17.9
  RBC, Normal | 67.0 | 65.8
  RBC, High | 17.7 | 16.3
  Neutrophils, Low: number analyzed (Participants) | 556 | 563
  Neutrophils, Low | 55.0 | 54.0
  Neutrophils, Normal: number analyzed (Participants) | 556 | 563
  Neutrophils, Normal | 44.6 | 45.6
  Neutrophils, High: number analyzed (Participants) | 556 | 563
  Neutrophils, High | 0.4 | 0.4
  Lymphocytes, Low: number analyzed (Participants) | 556 | 563
  Lymphocytes, Low | 1.8 | 3.7
  Lymphocytes, Normal: number analyzed (Participants) | 556 | 563
  Lymphocytes, Normal | 96.9 | 95.0
  Lymphocytes, High: number analyzed (Participants) | 556 | 563
  Lymphocytes, High | 1.3 | 1.2
  WBC, Low | 12.4 | 12.8
  WBC, Normal | 85.6 | 86.1
  WBC, High | 1.9 | 1.1
  Haemoglobin, Low | 23.6 | 25.7
  Haemoglobin, Normal | 74.6 | 73.4
  Haemoglobin, High | 1.8 | 1.0
  Platelets, Low | 1.9 | 1.7
  Platelets, Normal | 91.9 | 91.9
  Platelets, High | 6.2 | 6.3

12. Primary Outcome: Percentage of Subjects With Biochemical Laboratory Abnormalities
Description: Biochemical parameters assessed included: aminotransferase and creatinine. Reference range indicators used were: high, low, normal.
Time Frame: At Screening
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A Group | Placebo+GSK3390107A Group
Number analyzed (Participants) | 665 | 667
Percentage of participants
  Aminotransferase, Low | 4.7 | 5.1
  Aminotransferase, Normal | 92.9 | 93.3
  Aminotransferase, High | 2.4 | 1.6
  Creatinine, Low | 0 | 0.4
  Creatinine, Normal | 95.2 | 93.6
  Creatinine, High | 4.8 | 6.0

13. Primary Outcome: Percentage of Subjects With Biochemical Laboratory Abnormalities
Description: as for outcome 12
Time Frame: At Day 3
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A Group | Placebo+GSK3390107A Group
Number analyzed (Participants) | 660 | 662
Percentage of participants
  Aminotransferase, Low | 5.3 | 6.3
  Aminotransferase, Normal | 90.6 | 91.5
  Aminotransferase, High | 4.1 | 2.1
  Creatinine, Low | 0 | 0.2
  Creatinine, Normal | 94.4 | 93.8
  Creatinine, High | 5.6 | 6.0

14. Primary Outcome: Percentage of Subjects With Biochemical Laboratory Abnormalities
Description: as for outcome 12
Time Frame: At Day 6
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A Group | Placebo+GSK3390107A Group
Number analyzed (Participants) | 659 | 664
Percentage of participants
  Aminotransferase, Low | 5.6 | 6.9
  Aminotransferase, Normal | 91.8 | 89.5
  Aminotransferase, High | 2.6 | 3.6
  Creatinine, Low | 0 | 0.2
  Creatinine, Normal | 96.4 | 93.8
  Creatinine, High | 3.6 | 6.0

15. Primary Outcome: Percentage of Subjects With Biochemical Laboratory Abnormalities
Description: as for outcome 12
Time Frame: At Day 30
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A Group | Placebo+GSK3390107A Group
Number analyzed (Participants) | 659 | 663
Percentage of participants
  Aminotransferase, Low | 7.0 | 5.7
  Aminotransferase, Normal | 90.6 | 91.6
  Aminotransferase, High | 2.4 | 2.7
  Creatinine, Low | 0.2 | 0.3
  Creatinine, Normal | 93.8 | 93.5
  Creatinine, High | 6.1 | 6.2

16. Primary Outcome: Percentage of Subjects With Biochemical Laboratory Abnormalities
Description: as for outcome 12
Time Frame: At Month 6
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A Group | Placebo+GSK3390107A Group
Number analyzed (Participants) | 649 | 646
Percentage of participants
  Aminotransferase, Low | 6.5 | 6.2
  Aminotransferase, Normal | 91.8 | 90.4
  Aminotransferase, High | 1.7 | 3.4
  Creatinine. Low | 6.2 | 7.1
  Creatinine, Normal | 92.9 | 92.1
  Creatinine, High | 0.9 | 0.8

17. Primary Outcome: Percentage of Subjects With Biochemical Laboratory Abnormalities
Description: as for outcome 12
Time Frame: At Month 6 + 6 Days
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A Group | Placebo+GSK3390107A Group
Number analyzed (Participants) | 0 | 619
Percentage of participants
  Aminotransferase, Low |  | 6.1
  Aminotransferase, Normal |  | 91.3
  Aminotransferase, High |  | 2.6
  Creatinine, Low |  | 6.6
  Creatinine, Normal |  | 91.9
  Creatinine, High |  | 1.5

18. Primary Outcome: Percentage of Subjects With Biochemical Laboratory Abnormalities
Description: as for outcome 12
Time Frame: At Month 6 + 30 Days
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A Group | Placebo+GSK3390107A Group
Number analyzed (Participants) | 0 | 616
Percentage of participants
  Aminotransferase, Low |  | 4.2
  Aminotransferase, Normal |  | 93.5
  Aminotransferase, High |  | 2.3
  Creatinine, Low |  | 8.0
  Creatinine, Normal |  | 91.1
  Creatinine, High |  | 1.0

19. Primary Outcome: Percentage of Subjects With Biochemical Laboratory Abnormalities
Description: as for outcome 12
Time Frame: At Month 12
Population: as for outcome 11
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A Group | Placebo+GSK3390107A Group
Number analyzed (Participants) | 627 | 631
Percentage of participants
  Aminotransferase, Low | 6.9 | 6.7
  Aminotransferase, Normal | 90.7 | 89.7
  Aminotransferase, High | 2.4 | 3.6
  Creatinine, Low | 3.5 | 4.8
  Creatinine, Normal | 93.9 | 93.3
  Creatinine, High | 2.6 | 1.9

20. Primary Outcome: Number of Subjects With Adverse Events of Specific Interest (AESI)
Description: AESI included clinical symptoms of thrombocytopenia.
Time Frame: During the 7-Day (Days 0-6) post-vaccination period
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3390107A Group | Placebo+GSK3390107A Group
Number analyzed (Participants) | 749 | 751
Participants | 0 | 0

21. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (up to Month 12)
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3390107A Group | Placebo+GSK3390107A Group
Number analyzed (Participants) | 1509 | 1504
Participants | 11 | 18

22. Secondary Outcome: Concentrations of Anti-glycoprotein Ebola Zaire Virus (Anti-GP EBOV)
Description: Anti-GP EBOV antibody concentrations were measured by Enzyme-Linked Immunosorbent Assay (ELISA), presented as geometric mean concentrations (GMC), and expressed in ELISA units per milliliter (EU/mL).
Time Frame: At Day 0, Day 30, Month 6 and Month 12
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity - AE and Humoral Immunity Sub-cohort, which included all evaluable subjects for whom data concerning immunogenicity outcome measure were available.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | GSK3390107A Group | Placebo+GSK3390107A Group
Number analyzed (Participants) | 738 | 733
EU/mL
  Anti-GP EBOV, Day 0 | 31.961 [29.401 to 34.745] | 31.954 [29.405 to 34.724]
  Anti-GP EBOV, Day 30 | 900.025 [823.688 to 983.437] | 34.844 [31.864 to 38.103]
  Anti-GP EBOV, Month 6 | 458.649 [428.628 to 490.771] | 26.535 [24.732 to 28.471]
  Anti-GP EBOV, Month 12: number analyzed (Participants) | 738 | 0
  Anti-GP EBOV, Month 12 | 432.145 [401.725 to 464.869] |

23. Secondary Outcome: Percentage of Seronegative/Seropositive Subjects for Anti-GP EBOV Antibodies
Description: A seronegative subject (S-) is a subject whose titer is below (<) 36.11 EU/mL. A seropositive subject (S+) is a subject whose titer is greater than or equal to (≥) 36.11 EU/mL.
Time Frame: At Day 0, Day 30, Month 6 and Month 12
Population: as for outcome 22
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A Group | Placebo+GSK3390107A Group
Number analyzed (Participants) | 738 | 733
Percentage of participants
  Anti-GP EBOV, Day 0, S- | 74.8 | 74.9
  Anti-GP EBOV, Day 0, S+ | 25.2 | 25.1
  Anti-GP EBOV, Day 30, S-: number analyzed (Participants) | 731 | 726
  Anti-GP EBOV, Day 30, S- | 2.6 | 72.0
  Anti-GP EBOV, Day 30, S+: number analyzed (Participants) | 731 | 726
  Anti-GP EBOV, Day 30, S+ | 97.4 | 28.0
  Anti-GP EBOV, Month 6, S-: number analyzed (Participants) | 721 | 701
  Anti-GP EBOV, Month 6, S- | 0.7 | 81.9
  Anti-GP EBOV, Month 6, S+: number analyzed (Participants) | 721 | 701
  Anti-GP EBOV, Month 6, S+ | 99.3 | 18.1
  Anti-GP EBOV, Month 12, S-: number analyzed (Participants) | 693 | 0
  Anti-GP EBOV, Month 12, S- | 0.9 |
  Anti-GP EBOV, Month 12, S+: number analyzed (Participants) | 693 | 0
  Anti-GP EBOV, Month 12, S+ | 99.1 |

ADVERSE EVENTS:
Time Frame: Solicited and unsolicited adverse events: during the 30-day (Days 0-29) post-vaccination period; SAEs: up to study end (Month 12).
Description: Solicited and unsolicited AEs were collected only for subjects from the TVc- AEs and humoral immunity Sub-cohort, consisting of approximately 750 subjects per group, while SAEs were collected for all subjects included in the Total Vaccinated cohort (i.e. 3013).
Arm/Group | GSK3390107A Group | Placebo+GSK3390107A Group
All-Cause Mortality (participants affected / at risk) | 1/1509 | 2/1504
Serious Adverse Events (participants affected / at risk) | 11/1509 | 18/1504
Other Adverse Events (participants affected / at risk) | 530/749 | 230/751
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3390107A Group (N=1509) | Placebo+GSK3390107A Group (N=1504)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Malaria (Infections and infestations) | 2 (2) | 2 (2)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Snake bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
Face presentation (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Macrosomia (General disorders) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bladder outlet Obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3390107A Group (N=749) | Placebo+GSK3390107A Group (N=751)
Pain (General disorders) | 356 (680) | 60 (86)
Fatigue (General disorders) | 284 (448) | 94 (179)
Pyrexia (General disorders) | 106 (124) | 25 (30)
Headache (Nervous system disorders) | 345 (570) | 136 (249)
Gastrointestinal disorder (Gastrointestinal disorders) | 73 (125) | 49 (93)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.